CLINICAL TRIAL: NCT02666612
Title: Measurement and Characterization of Circulating Endothelial Cells or Circulating Tumor Cells or Circulating DNA in Adult Patients With Metastatic Cancer
Acronym: Liquid Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-A00585-50; 2008/1370 (Other: CSET number)
Record Dates: First submitted 2015-08-12; First posted 2016-01-28 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Cancer
Keywords: Patients
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with metastatic cancer (Other)
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples

SUMMARY:
Monitoring of circulating endothelial cells (CEC and mature cells called progenitors called CEP) or circulating tumor cells (CTC) in adult patients with metastatic cancer, possibly treated with targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic solid tumor
* Age> 18 years
* Signed consent

Exclusion Criteria:

* Patients with diseases associated with vascular lesions known.
* Patients protected by law, in accordance with Articles L1121-5 to L1121-8 of the Code of Public Health.
* Mental pathology that can interfere with the proper conduct of the study.
* Refusal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2240 (Estimated)
Dates: Start 2008-08 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Measurement and characterization of CEC and CEP and circulaing DNA rate using flow cytometry | up to 2 years
  Measurement and characterization of initial CEC and CEP circulaing DNA and their evolution under treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Charles Soria, MD-PhD, Study Chair — Gustave Roussy Cancer Campus
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France